CLINICAL TRIAL: NCT02820922
Title: Anesthetic Techniques for Emergency Orthopedic Surgery
Brief Title: Anesthesia for Emergency Orthopedic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Havva Sayhan, Assistant Professor, Sakarya University
Other Study IDs: Sakarya University
Record Dates: First submitted 2016-06-24; First posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Anesthesia
Keywords: Emergency orthopedic surgery; anesthesia; general anesthesia; regional anesthesia
MeSH Terms: interventions — Orthopedic Procedures; Anesthesia, Conduction; Anesthesia, General

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Orthopedic emergency surgery: Patients of all ages who have undergone emergency orthopedic surgery The analysis of medical data with regard to age, sex, the American Society of Anesthesiologists (ASA) score, anaesthesia technique, comorbidities, surgery diagnosis, length of surgery, complications and admission to intensive care unit after surgery
  Interventions: Procedure: Orthopedic

INTERVENTIONS:
Procedure: Orthopedic — anesthesia techniques with regard to age, sex, ASA score, anaesthesia technique, comorbidities, surgery diagnosis, length of surgery, complications and admission to intensive care unit after surgery
  Other Names: regional anesthesia; sedation; general anesthesia

SUMMARY:
The aim of this retrospective study is to evaluate the preferred anaesthesia techniques in our clinic for emergency orthopedic surgery at a 1 year period.

DETAILED DESCRIPTION:
This retrospective study included patients of all ages who have undergone emergency orthopedic surgery between January 2015 and December 2015 after approval of the research ethics committee. Medical record forms and electronic medical record system of the hospital were used in the analysis of medical data with regard to age, sex, ASA score, anaesthesia technique, comorbidities, surgery diagnosis, length of surgery, complications and admission to intensive care unit after surgery.

ELIGIBILITY:
Inclusion Criteria:

* all patients who had orthopedic emergency surgery

Exclusion Criteria:

* involvement of incomplete data collection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all age groups who administered for orthopedic emergency surgery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-02 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with preferred anesthesia technique for orthopedic emergency surgery assessed by Statistical Package for the Social Sciences (SPSS) v22.0 | 1 year
  Statistical assessment would be carried out with regard to anesthesia technique. Outcome measures the number of patients with demographic data arrive at orthopedic emergency service. Results will be helpful on preferred anesthesia technique at orthopedic emergency surgery in our clinic.

SECONDARY OUTCOMES:
Assessment of ages and anesthesia technique relation on orthopedic emergency surgery by SPSS v22.0 | 3 months
  Age is a factor that make changes relevant to anesthesia. The study analyze the influence of age on anesthesia technique at orthopedic emergency surgery.
Assessment of orthopedic surgery type and anesthesia relation on orthopedic emergency surgery by SPSS v22.0 | 3 months
  Statistical evaluation of orthopedic surgery type relevant to anesthesia. The study analyze the influence of surgery type on preferred anesthesia technique at our hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Ali F Erdem, Prof, Study Chair — Sakarya University
Locations (1):
- Sakarya University Research and Training Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark L, Robinson M, Varbanova M. Role of regional anesthesia in orthopedic trauma. Anesthesiol Clin. 2014 Dec;32(4):789-808. doi: 10.1016/j.anclin.2014.08.002. Epub 2014 Nov 25. PMID 25453662
- [Background] Stundner O, Ortmaier R, Memtsoudis SG. Which outcomes related to regional anesthesia are most important for orthopedic surgery patients? Anesthesiol Clin. 2014 Dec;32(4):809-21. doi: 10.1016/j.anclin.2014.08.003. Epub 2014 Nov 25. PMID 25453663
- [Background] Campbell VL. Anesthetic protocols for common emergencies. Vet Clin North Am Small Anim Pract. 2005 Mar;35(2):435-53. doi: 10.1016/j.cvsm.2004.10.005. PMID 15698919
- See also: book chapter link — http://cdn.intechopen.com/pdfs/31589.pdf
- See also: book — http://link.springer.com/chapter/10.1007%2F88-470-0407-1_61